CLINICAL TRIAL: NCT04937127
Title: Efficacité du E-learning et du Jeu de rôle Pour la Formation Des Soignants Des EHPAD à l'Accompagnement de l'Agitation Dans Les Maladies neurodégénératives : Essai randomisé en Cluster
Brief Title: Efficiency of E-learning and Role-playing for the Training of Nursing Home Caregivers in the Support of Agitation in Neurodegenerative Diseases
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR200087 (I-LEARN)
Record Dates: First submitted 2021-06-08; First posted 2021-06-23 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Neuro-Degenerative Disease
Keywords: agitation; dependent elderly people; psycho-behavioral disorders; nursing home
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: The experimental group will be made up of patients from nursing homes whose carers have received I-Learn training.
  Interventions: Behavioral: I-LEARN training; Other: usual care
- Control Group: The control group will consist of nursing homes patients whose caregivers have not received I-Learn training and will continue their usual care, regardless of the practices already implemented.
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: I-LEARN training — Training of psycho-behavorial disorders care in neurodegenerative diseases: including a theoretical part in e-learning and a practical part
  Groups: Experimental Group
Other: usual care — usual care

SUMMARY:
This study will investigate the effects of "I-Learn cognition and behaviour" training in the care in agitation in patients with neurodegenerative diseases. This training for caregivers, aims to reduce agitation and psycho-behavioral disorders of patients living in nursing home. In addition, amount of psychotropic drugs prescribed, as well as the number of hospitalizations during the study will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Neurocognitive Disorder according to DSM 5
* With agitation and NPI agitation item score of 4 or more (frequency X severity)
* Information and verification of the non-opposition of the patient and his guardian / curator if he is under legal protection.

Exclusion Criteria:

* Patient under court protection
* Inability to understand the French language
* Patient whose state of health is not stabilised at the time of inclusion and/or in palliative care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dependent elderly people with a neurodegenerative disease
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Measurement of agitation of patients in the nursing home | Baseline
  Assessment of agitation using the Cohen-Mansfield Agitation Inventory (CMAI, 1989) by asking caregivers about the patients' behaviour.
  The minimum value is 0 and the maximum value is 203. the higher the score, the more intense the agitation
Measurement of agitation of patients in the nursing home | 3 months
  Assessment of agitation using the Cohen-Mansfield Agitation Inventory (CMAI, 1989) by asking caregivers about the patients' behaviour.
  The minimum value is 0 and the maximum value is 203. the higher the score, the more intense the agitation
Measurement of agitation of patients in the nursing home | 6 months
  Assessment of agitation using the Cohen-Mansfield Agitation Inventory (CMAI, 1989) by asking caregivers about the patients' behaviour.
  The minimum value is 0 and the maximum value is 203. the higher the score, the more intense the agitation
Measurement of agitation of patients in the nursing home | 9 months
  Assessment of agitation using the Cohen-Mansfield Agitation Inventory (CMAI, 1989) by asking caregivers about the patients' behaviour.
  The minimum value is 0 and the maximum value is 203. the higher the score, the more intense the agitation

SECONDARY OUTCOMES:
Frequency and severity of Psychobehavioural Symptoms associated with Dementia | Baseline, 3 months, 6 months and 9 months
  Assessment using the Neuro Psychiatric Inventory, care team version (NPI-ES, 2000). 10 behavioural domains and 2 neurovegetative variables are considered. item score = frequency x severity frequency minimum = 1 and maximum = 4 severity minimum = 1 and maximum = 3 A score above 2 is pathological
Quality of life of patients | Baseline, 3 months, 6 months and 9 months
  Assessment using the Quality of Life-Alzheimer's Disease (QOL-AD, 2009) 13 questions focus on the patient's quality of life. the patient's current quality of life in each domain is assessed by choosing one of the following four words: poor, fair, good, excellent.
Impact of I-Learn on psychotropic drug prescriptions | Baseline, 3 months, 6 months and 9 months
  Changes in the prescriptions given to patients in terms of psychotropic drugs (addition or withdrawal of a neuroleptic, antidepressant, anxiolytic, etc.)
Impact of I-Learn on psychotropic drug prescriptions | Baseline, 3 months, 6 months and 9 months
  Changes in the prescriptions given to patients in terms of dosage (increase/decrease of the daily dose)
Impact of I-Learn training on hospital admissions | 3 months, 6 months and 9 months
  number of transfers to acute or emergency departments
Impact of I-Learn training on hospital admissions | 3 months, 6 months and 9 months
  reasons for hospitalisation
Impact of Psychobehavioural Symptoms Associated with Dementia on the professional practice of health care teams | Baseline, 3 months, 6 months and 9 months
  Assessment using the Neuro Psychiatric Inventory, care team version (NPI-ES, 2000) 10 behavioural domains and 2 neurovegetative variables are considered. item score = frequency x severity fequency minimum = 1 and maximum = 4 severity minimum = 1 and maximum = 3 A score above 2 is pathological
Caregiver burnout at work | Baseline, 6 months and 9 months
  Assessment using the Maslach Burnout Inventory (MBI, 1986) 22 items For each item, the minimum value is 0 and the maximum value is 6 BURNOUT Questions 1.2.3.6.8.13.14.16.20 Degree of burn out Total below 17 = low Total between 18 and 29 = moderate Total above 30 = high
  DEPERSONALISATION Questions 5.10.11.15.22 Degree of burn out Total below 5 = low Total between 6 and 11 = moderate Total above 12 = high
  PERSONAL FULFILMENT Questions 4.7.9.12.17.18.19.21 Degree of burn out Total above 40 = low Total between 34 and 39 = moderate Total below 33 = high
  Moderate or even high scores are a sign of latent burnout that is taking hold.

CONTACTS AND LOCATIONS:
Overall Officials: Céline LOURDEL, Principal Investigator — University Hospital, Tours
Locations (7):
- France (7):
  - EHPAD Résidence du Prévot, Châteaugiron
  - Maison Saint Michel, Liffré
  - EHPAD La Bourdaisière, Montlouis-sur-Loire
  - Résidence Père Brottier, Pléchâtel
  - EHPAD Le Clos Saint-Vincent, Rochecorbon
  - EHPAD Montconseil, Tours
  - EHPAD La Source, Tours

IPD SHARING:
Plan to Share IPD: Undecided